CLINICAL TRIAL: NCT03159962
Title: Mandibular Response After Rapid Maxillary Expansion in Class II Growing Patients: a Pilot Randomized Controlled Trial
Brief Title: Mandibular Response After Maxillary Orthopedic Expansion in Class II Growing Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Lione, Principal Investigator, Research Fellow, Department of Clinical Sciences and Translational Medicine, University of Rome "Tor Vergata," Rome, Italy, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130/14
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Malocclusion, Angle Class II; Malocclusion
Keywords: Rapid maxillary expansion; Mandibular response; Class II malocclusion; Growing subjects
MeSH Terms: conditions — Malocclusion, Angle Class II; Malocclusion; Overbite

STUDY DESIGN:
Intervention Model Description: prospective 3-arm parallel group randomized clinical trial with a 1:1:1 allocation ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treated Group 1 (Active Comparator): Patient treated with bonded RME (Rapid Maxillary Expander) with a 13-mm screw. The acrylic splints of the bonded expander extended from the first deciduous molars through the first permanent molars.
  Interventions: Device: Bonded RME (Rapid Maxillary Expander) appliance
- Treated Group 2 (Active Comparator): Patients treated with banded RME (Rapid Maxillary Expander) in the form of a butterfly palatal expander with a 13-mm screw cemented through bands on the second deciduous upper molars.
  Interventions: Device: Banded RME (Rapid Maxillary Expander) appliance
- Untreated Control Group (No Intervention): Matched untreated Class II control group prospectively evaluated after one year

INTERVENTIONS:
Device: Bonded RME (Rapid Maxillary Expander) appliance — The expansion screw was activated 1 quarter of a turn per day (0.25 mm per turn) until the palatal cusps of the maxillary posterior teeth approximated the lingual cusps of the mandibular posterior teeth.
  The expander was kept in place as a passive retainer for 8 months. After expander removal, patients were followed without performing any additional treatment for 4 months.
  Arms: Treated Group 1
Device: Banded RME (Rapid Maxillary Expander) appliance — The expansion screw was activated 1 quarter of a turn per day (0.25 mm per turn) until the palatal cusps of the maxillary posterior teeth approximated the lingual cusps of the mandibular posterior teeth.
  The expander was kept in place as a passive retainer for 8 months. After expander removal, patients were followed without performing any additional treatment for 4 months.
  Arms: Treated Group 2

SUMMARY:
the effectiveness of RME (Rapid Maxillary Expander) on the sagittal dental or skeletal parameters is still controversial because very little has been written regarding the behavior of antero-posterior mandibular changes in Class II growing subjects who underwent RME as the phase 1 treatment intervention. The reported significant occlusal improvement could be attributed to other reasons, ie, skeletal growth or the use of additional appliances during transition from mixed to permanent dentition. Moreover, the majority of the studies show some limits: they are not randomized, they are not prospective, and they have no control group or they use patients from growth studies as a source for the control group. The primary objective of the present investigation was to conduct a pilot randomized controlled trial (RCT) evaluating the changes in the antero-posterior mandibular position induced by bonded or banded RMEs compared with an untreated Class II control group

DETAILED DESCRIPTION:
Class II malocclusions are commonly observed in orthodontic patients. During treatment planning among the several dento-skeletal pattern combinations of Class II malocclusion, it is important to consider the maxillary transverse deficiency, which is often overlooked.

it has been showed showed an underlying posterior interarch transverse discrepancy of 3 to 5 mm in subjects in early mixed dentition with Class II malocclusions without posterior crossbites in centric occlusion. When these Class II patients are asked to posture their lower jaw forward in a Class I molar relationship, this transverse discrepancy (ie, maxillary constriction) can be observed clinically. It was postulated that in these subjects the mandible is kept in a distal position relative to centric relation because the constricted maxilla is holding it back. The presence of a primitive transverse discrepancy between the dental arches induces a backward position of the mandible, as the occlusal goal is to obtain the highest number of functional contacts.

As reported by several authors, widening the maxilla with rapid maxillary expansion often leads to spontaneous forward posturing of the mandible during the retention period. The orthopedic expansion removes occlusal interferences, allowing the mandible to posture forward, thus improving the sagittal relationships. The mandibular arch acts as a ''foot'' that moves forward after the ''shoe'' is widened.

However, the effectiveness of RME on the sagittal dental or skeletal parameters is still controversial because very little has been written regarding the behavior of antero-posterior mandibular changes in Class II growing subjects who underwent RME as the phase 1 treatment intervention. The reported significant occlusal improvement could be attributed to other reasons, ie, skeletal growth or the use of additional appliances during transition from mixed to permanent dentition. Moreover, the majority of the studies show some limits: they are not randomized, they are not prospective, and they have no control group or they use patients from growth studies as a source for the control group.

Considering that it was not possible to estimate from previous studies the standard deviation to be used for sample size calculation of the main trial with special regards to type of intervention and observation intervals, the primary objective of the present investigation was to conduct a pilot randomized controlled trial (RCT) evaluating the changes in the antero-posterior mandibular position induced by bonded or banded RMEs compared with an untreated Class II control group.

To evaluate the sagittal mandibular response induced by RME therapy in mixed dentition patients with Class II malocclusion, comparing the effects of bonded RME and banded RME with a matched untreated Class II control group

This is a single center, prospective 3-arm parallel group randomized clinical trial with a 1:1:1allocation ratio. 30 (thirty) of subjects are planned. Each subject in the treated groups will be treated with a Rapid Maxillary Expander (RME), bonded or banded respectively. Subjects will be assigned to the groups in random order. Evaluations will be taken at baseline and at the end of the retention period/follow up (for a total of 12 months). Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Allocation of patients to the three groups in a 1:1:1 ratio was determined by a computer-generated randomization list using Rv.0.1 software and by a block size of 4. Then, the allocation information (randomization results) was concealed in opaque and sealed envelopes by the statistician.

The study was blinded in regard of the statistical analysis. Data were recorded and blinded for the statistician: blinding was obtained by eliminating from the elaboration file every reference to patient group assignment

To determine the reliability of the method 15 radiographs chosen at random were traced and digitized by the same investigator on 2 separate occasions at least one month apart. A paired t-test was used to compare the two measurements (systematic error). The magnitude of the random error was calculated by using the method of moment's estimator (MME). Exploratory statistics revealed that not all cephalometric variables were normally distributed (Kolmogorov-Smirnov test) with equality of variances (Levene's test).Kruskal-Wallis test or ANOVA with Tukey's post-hoc tests were used to compare the T2-T1 changes in the three groups. All changes were considered significant at P<0.05. All statistical computations were performed with Statistical Package for the Social Sciences software (Version 12, Chicago, IL)..

10 randomized subjects will be included in the treated group 1, 10 randomized patients will be included in the treated group 2 and 10 randomized patients will be used as untreated control group.

The baseline age was 8.1 ± 0.6 years (range 6.6-9.1 years).

Sample size for this pilot trial was calculated according to the method proposed by Whitehead et al. For a standardized effect size of 1 (a clinically relevant change of 2.0 mm with a combined Standard Deviation of 2.0 mm derived from Guest et al.) for the 8 primary outcome variable Pogonion to Nasion perpendicular, a sample size of 10 subjects per group was required for a Type I error rate of 5% and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* early mixed dentition with first molars fully erupted,
* Class II malocclusion (full-cusp or end-to-end molar relationships),
* negative posterior transverse interarch discrepancy ≥ 4 mm,
* Overjet ≥ 5 mm,
* and prepubertal stage of development (Cervical Stage 1 - Cervical Stage 2 in cervical vertebral maturation)

Exclusion Criteria:

* previous orthodontic treatment,
* extracted or congenitally missing teeth,
* craniofacial syndromes or clefts,
* use of additional orthodontic devices during the observation period

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mandibular displacement after RME appliance therapy (linear measurement in millimeters) when compared with a matched untreated control group | 12 months
  The primary outcome was the change in the position of point Pogonion to the Nasion perpendicular (Pg to N perp). The objective is to evaluate the changes in the sagittal mandibular position induced by bonded or banded RMEs compared with an untreated control group.
  For each treated patient, standard lateral cephalograms were obtained before treatment and after 1 year to evaluate the dento-skeletal changes. The Control Group was followed up without treatment for 1 year and had lateral cephalograms before and after a one-year interval.
  Cephalograms were scanned using a professional table scanner (Epson Perfection V700 Photo, CA, USA), with resolution set to 150 dots per inch (dpi) gray scale and were digitized by 1 investigator., followed by a customized digitization regimen and analysis (Viewbox 3.1; dHAL Software, Kifissia, Greece). All cephalograms were at a magnification of 0%. The examiner was blinded to the origin of the films and the group to which each subject belonged

SECONDARY OUTCOMES:
Occlusal improvement of Class II molar relationship after RME appliance therapy (linear measurement in millimeters) when compared with a matched untreated control group | 12 months
  The secondary outcome is to evaluate if maxillary expansion corrects or improves a Class II molar relationship (the mesiobuccal cusp of the maxillary permanent 1st molar must occlude in the embrasure between the mandibular 2nd premolar and the mandibular permanent 1st molar) when compared with an untreated control group. For each treated patient, lateral cephalograms were obtained before treatment and after 1 year to evaluate the dento-skeletal changes. Untreated patients had lateral cephalograms before and after a 1 year interval. Cephalograms were scanned using a professional table scanner (Epson Perfection V700 Photo, CA, USA), with resolution set to 150 dots per inch (dpi) gray scale and were digitized by 1 investigator., followed by a customized digitization regimen and analysis (Viewbox 3.1; dHAL Software, Kifissia, Greece). All cephalograms were at a magnification of 0%. The examiner was blinded to the origin of the films and the group to which each subject belonged
Treatment effects on vertical dimension (SN-Go Me; angular measurement) and on Gonial Angle (Ar-Go-Me, angular measurement) and vertical growth pattern after RME appliance therapy when compared with a matched untreated control group | 12 months
  The objective is to verify if the treatment determined a reduction of the facial divergency (SN-Go Me°) and of the gonial angle (Ar-Go-Me°) when both subjects, treated respectively with banded RME and bonded RME, are compared with untreated subjects.
  For each treated patient, standard lateral cephalograms were obtained before treatment and after 1 year to evaluate the dento-skeletal changes. The Control Group was followed up without treatment for 1 year and had lateral cephalograms before and after a one-year interval.
  Cephalograms were scanned using a professional table scanner (Epson Perfection V700 Photo, CA, USA), with resolution set to 150 dots per inch (dpi) gray scale and were digitized by 1 investigator., followed by a customized digitization regimen and analysis (Viewbox 3.1; dHAL Software, Kifissia, Greece). All cephalograms were at a magnification of 0%. The examiner was blinded to the origin of the films and the group to which each subject belonged

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Lione, Dentistry, Principal Investigator — Research Fellow, Department of Clinical Sciences and Translational Medicine, University of Rome "Tor Vergata," Rome, Italy, and research Fellow, Department of Dentistry, University Nostra Signora del Buon Consiglio, Tirana, Albania
Locations (1):
- University of Rome "Tor Vergata", Rome, Italy

IPD SHARING:
Plan to Share IPD: No
no individual participant data are to be shared

REFERENCES:
- [Background] McNamara JA Jr, Sigler LM, Franchi L, Guest SS, Baccetti T. Changes in occlusal relationships in mixed dentition patients treated with rapid maxillary expansion. A prospective clinical study. Angle Orthod. 2010 Mar;80(2):230-8. doi: 10.2319/040309-192.1. PMID 19905846
- [Result] Baratieri C, Alves M Jr, Bolognese AM, Nojima MC, Nojima LI. Changes in skeletal and dental relationship in Class II Division I malocclusion after rapid maxillary expansion: a prospective study. Dental Press J Orthod. 2014 May-Jun;19(3):75-81. doi: 10.1590/2176-9451.19.3.075-081.oar. PMID 25162569
- [Result] Baccetti T, Franchi L, McNamara JA Jr, Tollaro I. Early dentofacial features of Class II malocclusion: a longitudinal study from the deciduous through the mixed dentition. Am J Orthod Dentofacial Orthop. 1997 May;111(5):502-9. doi: 10.1016/s0889-5406(97)70287-7. PMID 9155809
- [Result] Tollaro I, Baccetti T, Franchi L, Tanasescu CD. Role of posterior transverse interarch discrepancy in Class II, Division 1 malocclusion during the mixed dentition phase. Am J Orthod Dentofacial Orthop. 1996 Oct;110(4):417-22. doi: 10.1016/s0889-5406(96)70045-8. PMID 8876494
- [Result] McNamara JA. Maxillary transverse deficiency. Am J Orthod Dentofacial Orthop. 2000 May;117(5):567-70. doi: 10.1016/s0889-5406(00)70202-2. No abstract available. PMID 10799117
- [Result] Guest SS, McNamara JA Jr, Baccetti T, Franchi L. Improving Class II malocclusion as a side-effect of rapid maxillary expansion: a prospective clinical study. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):582-91. doi: 10.1016/j.ajodo.2008.12.026. PMID 21055598
- [Result] Wendling LK, McNamara JA Jr, Franchi L, Baccetti T. A prospective study of the short-term treatment effects of the acrylic-splint rapid maxillary expander combined with the lower Schwarz appliance. Angle Orthod. 2005 Jan;75(1):7-14. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15747809
- [Result] Feres MF, Raza H, Alhadlaq A, El-Bialy T. Rapid maxillary expansion effects in Class II malocclusion: a systematic review. Angle Orthod. 2015 Nov;85(6):1070-9. doi: 10.2319/102514-768.1. PMID 26516713
- [Result] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Result] Springate SD. The effect of sample size and bias on the reliability of estimates of error: a comparative study of Dahlberg's formula. Eur J Orthod. 2012 Apr;34(2):158-63. doi: 10.1093/ejo/cjr010. Epub 2011 Mar 29. PMID 21447784
- [Result] Baratieri C, Alves M Jr, Sant'anna EF, Nojima Mda C, Nojima LI. 3D mandibular positioning after rapid maxillary expansion in Class II malocclusion. Braz Dent J. 2011;22(5):428-34. doi: 10.1590/s0103-64402011000500014. PMID 22011901
- [Result] Volk T, Sadowsky C, Begole EA, Boice P. Rapid palatal expansion for spontaneous Class II correction. Am J Orthod Dentofacial Orthop. 2010 Mar;137(3):310-5. doi: 10.1016/j.ajodo.2008.05.017. PMID 20197166
- [Result] Schulz SO, McNamara JA Jr, Baccetti T, Franchi L. Treatment effects of bonded RME and vertical-pull chincup followed by fixed appliance in patients with increased vertical dimension. Am J Orthod Dentofacial Orthop. 2005 Sep;128(3):326-36. doi: 10.1016/j.ajodo.2004.03.039. PMID 16168329
- [Result] Asanza S, Cisneros GJ, Nieberg LG. Comparison of Hyrax and bonded expansion appliances. Angle Orthod. 1997;67(1):15-22. doi: 10.1043/0003-3219(1997)0672.3.CO;2. PMID 9046395
- [Derived] Lione R, Brunelli V, Franchi L, Pavoni C, Quiroga Souki B, Cozza P. Mandibular response after rapid maxillary expansion in class II growing patients: a pilot randomized controlled trial. Prog Orthod. 2017 Nov 6;18(1):36. doi: 10.1186/s40510-017-0189-6. PMID 29105023